CLINICAL TRIAL: NCT06113640
Title: Clinical Study to Investigate the Possible Efficacy and Safety of Montleukast in Parkinson Disease
Brief Title: Montelukast in Parkinson Disease
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mostafa Bahaa (Other)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Teaching assisstant, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4789
Record Dates: First submitted 2023-10-28; First posted 2023-11-02 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination; montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Control group (Levo-dopa group, n =30) who received levodopa/carbidopa (250/25 mg) three times daily for 12 months
  Interventions: Drug: levodopa-carbidopa
- Montelukast group (Active Comparator): who received levodopa/carbidopa (250/25 mg) three times daily plus Montelukast 10 mg once daily for 12 months
  Interventions: Drug: levodopa-carbidopa; Drug: Montelukast

INTERVENTIONS:
Drug: levodopa-carbidopa — Carbidopa/levodopa, also known as levocarb and co-careldopa, is the combination of the two medications carbidopa and levodopa. It is primarily used to manage the symptoms of Parkinson's disease
Drug: Montelukast — Montelukast and other CysLT1 antagonists are currently used as an adjuvant therapy for children and adults suffering from asthma. Other indications have been proposed and most evidence exists for the use of montelukast to treat allergic rhinitis, but its use in other inflammatory conditions, such as atherosclerosis and chronic obstructive pulmonary disease, have also been suggested.
  Arms: Montelukast group

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disorder after Alzheimer's disease (AD). Clinical manifestations of PD can vary, but a formal diagnosis relies on the presence of bradykinesia with rigidity and/or rest tremor according to Movement Disorder Society (MDS) criteria for PD. Non-motor symptoms, such as hyposmia, constipation, depression, and rapid eye movement (REM) sleep behavior disorder, are common and can in many cases manifest before classical motor symptoms. In later years, more emphasis has been put on non-motor symptoms, especially in the early stages of PD and which is evident in the proposed prodromal PD criterion by MDS.

DETAILED DESCRIPTION:
Leukotrienes are along with prostaglandins, lipoxins, and thromboxanes included in a group of long-chain fatty acids known as eicosanoids. They are known to play important parts in the inflammatory response such as leukocyte chemotaxis, vascular leakage, and astrocyte proliferation, and were first described by Bengt Samuelsson and colleagues in 1983. Leukotrienes (LT) are synthesized from free arachidonic acid (AA) by the enzyme 5-lipoxygenase (5-LOX) into LTA4, which is then further metabolized into LTB4, C4, D4, and E4. LTC4, D4, and E4 are grouped by their molecule structure to form the cysteinyl leukotrienes and they mainly activate two receptors, CysLT1 and CysLT2. CysLT1 is a Gq/11 family G-protein-coupled receptor with signaling through phospholipase C and Ca2+ mobilization

ELIGIBILITY:
Inclusion Criteria:

- Age ≥ 18 years Both male and female will be included Negative pregnancy test and effective contraception. Diagnosed Parkinson's disease patient taking Levodopa

Exclusion Criteria:

- Secondary causes of parkinsonism Patients taking anti-inflammatory drugs Atypical parkinsonian syndromes Prior stereotaxic surgery for Parkinson's disease Pregnancy and lactation Suffering from active malignancy Addiction to alcohol and / or drugs Known allergy to the studied medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in unified parkison disease rating scale | 12 months
  The Unified Parkinson's Disease Rating Scale (UPDRS) is the most widely applied rating instrument for Parkinson disease (PD). The Total UPDRS score includes 31 items contributing to three subscales: (I) Mentation, Behavior, and Mood; (II) Activities of Daily Living; and (III) Motor Examination

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Mansoura University, Al Mansurah, Egypt